CLINICAL TRIAL: NCT05939271
Title: Lower Extremity Amputations in Persons With Diabetes Mellitus in the Netherlands, a Retrospective Study Using an All-payer Claims Database
Brief Title: Lower Extremity Amputations in Persons With Diabetes Mellitus in the Netherlands
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Isala (Other); Innofeet (Unknown); Vektis health care information center (Unknown); National Institute for Public Health and the Environment (RIVM) (Other Government)
Responsible Party: Sponsor
Other Study IDs: Dude 6-449
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Lower Extremity Amputations; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- persons with DM who underwent a lower extremity amputation
  Interventions: Procedure: lower extremity amputation
- persons with DM who did not underwent a lower extremity amputation
- persons without DM who underwent a lower extremity amputation
  Interventions: Procedure: lower extremity amputation

INTERVENTIONS:
Procedure: lower extremity amputation — persons are defined as having a lower extremity amputation when an operation with removal of an extremity below the hips took place.
  To identify those people with diabetes who underwent amputation, the following DBC's claims were extracted from the system: "038590; amputation upper leg", "038690; amputation lower leg", "038691; exarticulation of the lower leg", 038790; amputation of the tarsus", "038791; amputation or exarticulation of a toe", "038793; exarticulation of the foot", "038794; Chopart exarticulation, Lisfranc, respectively trans metatarsal amputation". Amputations were categorized into minor (038790, 038791, 038793, 038794) and major (038590, 038690,038691) amputations
  Groups: persons with DM who underwent a lower extremity amputation; persons without DM who underwent a lower extremity amputation

SUMMARY:
This is a retrospective, observational study based on an all-payer claims database (APCD) in the period 2011 to 2020) managed by the Vektis Health Care Information Center. In 2006, Vektis was established by Dutch health insurers aiming to combine and interpret reimbursement data and enable the main players in the Dutch healthcare market to base decisions and policy on reliable, essential, and timely information. Vektis receives data from all Dutch health care insurers. The APCD covers health care claims of 99.9% of the Dutch population. This study is part of the DUtch Diabetes Estimates (DUDE) initiative. We aim to perform different predefined analyses with the available data:

* What is the incident amputation rate in persons with and without DM in the Netherlands in the period 2011-2020?
* What defines persons with DM who need an amputation as compared to matched persons with DM but without an amputation in 2016, both in aspects of health care use and costs?
* What defines persons with DM who need an amputation as compared to matched persons without DM with an amputation?
* Does Social Economic Status (SES) play a role in amputation incidence and level, or on longer term outcome in persons with DM in the Netherlands?
* Does the presence of a formal multidisciplinary foot clinic / team in a hospital make a difference, especially when comparing previous and actual macrovascular complication rates?

ELIGIBILITY:
Inclusion Criteria:

* All persons aged ≥ 18 years, diagnosed with type 1 DM (T1DM) or type 2 DM (T2DM) identified in the Vektis data met the inclusion criteria

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons aged ≥ 18 years, diagnosed with type 1 DM (T1DM) or type 2 DM (T2DM) and matching persons without diabetes.
Sampling Method: Probability Sample
Enrollment: 2808 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
- What is the incident amputation rate in persons with and without DM in the Netherlands in the period 2011-2020? | dec 23

SECONDARY OUTCOMES:
- What defines persons with DM who need an amputation as compared to matched persons with DM but without an amputation in 2016, both in aspects of health care use and costs? | dec 23
- What defines persons with DM who need an amputation as compared to matched persons without DM with an amputation? | dec23
- Does Social Economic Status (SES) play a role in amputation incidence and level, or on longer term outcome in persons with DM in the Netherlands? | dec 23
- Does the presence of a formal multidisciplinary foot clinic / team in a hospital make a difference, especially when comparing previous and actual macrovascular complication rates? | dec24

CONTACTS AND LOCATIONS:
Locations (1):
- L. Rosien, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No
The datasets are not publicly available, as formal consent from the Dutch health insurers is needed to gain access to these files. Data could made available from Vektis Health Care Information Center upon reasonable request and with formal consent of the Dutch health insurers.